CLINICAL TRIAL: NCT03841591
Title: Maternal Weight Gain in Gestational Diabetes Controlled by Metformin Versus Insulin: A Randomized Controlled Trial
Brief Title: Maternal Weight Gain in Gestational Diabetes Controlled by Metformin Versus Insulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sinaa Hamdy Abo ElWafa, Resident of O&G, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MatWt-GDM
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Insulin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin Group (Active Comparator): This includes women with GDM allocated to receive insulin treatment. Starting dose will be 30unit (20 unit intermediate dose + 10 unit rapid acting insulin) in the morning and before breakfast). In the 2nd trimester, we will start with half of the previous dose and if post dinner glucose level remain elevated additional injection of rapid acting insulin will be given just prior to dinner. If fasting glucose is elevated, intermediate acting insulin can be given along with the dinner dose of rapid acting insulin.
  Interventions: Drug: Insulin; Other: Assessment of weight gain
- Metformin Group (Active Comparator): This includes women with GDM allocated to receive metformin treatment. They will receive an initial metformin dose of 500 mg once or twice daily (according to initial blood glucose level) with food and increased 500 mg every one or two weeks toward targets or up to a maximum daily dose of 2500 mg divided doses with each meal.
  Interventions: Drug: Metformin; Other: Assessment of weight gain

INTERVENTIONS:
Drug: Insulin — Women with GDM will receive insulin and tailored according to their blood glucose levels to achieve glycemic control. Starting dose will be 30unit (20 unit intermediate dose + 10 unit rapid acting insulin) in the morning and before breakfast). In the 2nd trimester, we will start with half of the previous dose and if post dinner glucose level remain elevated additional injection of rapid acting insulin will be given just prior to dinner. If fasting glucose is elevated, intermediate acting insulin can be given along with the dinner dose of rapid acting insulin.
  Arms: Insulin Group
Drug: Metformin — Women with GDM will receive metformin and tailored according to their blood glucose levels to achieve glycemic control. They will receive an initial metformin dose of 500 mg once or twice daily (according to initial blood glucose level) with food and increased 500 mg every one or two weeks toward targets or up to a maximum daily dose of 2500 mg divided doses with each meal.
  Other Names: Cidophage
  Arms: Metformin Group
Other: Assessment of weight gain — Body weight will be measured monthly from the start of treatment till delivery.

SUMMARY:
Insulin has many disadvantages for mothers with GDM including the need to give injections, frequent daily testing for monitoring, and risks of hypoglycemia, increase in appetite, weight gain and high cost. Metformin, an oral biguanide, may be a more logical alternative to insulin for women with GDM who are unable to cope with the increasing insulin resistance of pregnancy.

This study aim to compare maternal weight gain during pregnancy in women with gestational diabetes, treated by insulin versus metformin.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged (19-35) years
* BMI 18-30 kg/m2
* Gestational age >24 weeks
* Singleton pregnancy
* Gestational diabetes mellitus with failure to achieve adequate glucose control on diet therapy alone (FBG > 105) OR patients with gestational diabetes who are controlled with either metformin alone or insulin alone.

Exclusion Criteria:

* Pregnant women with preexisting diabetes mellitus
* Women who have contraindication to take metformin e.g.: impaired renal function, hepatic cirrhosis, hepatitis).
* Patients with other medical disorders that could affect perinatal outcome (e.g., hypertension, SLE etc).
* Fetal anomalies identified on ultrasound prior to initiation of therapy.
* Patients who refused to participate

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Rate of maternal weight gain per week | 4 months
  Maternal weight (in grams) will be measured monthly. Difference in measured weight between starting treatment and delivery will be divided by the number of weeks.

SECONDARY OUTCOMES:
1-min APGAR score | 1 minute
  APGAR score at minute 1 after delivery
5-min APGAR score | 5 minutes
  APGAR score at minute 5 after delivery
Incidence of neonatal hypoglycemia | 1 day
  Number of neonates with two or more neonatal glucose value <2.6 mmol per liter during the first day after delivery.
Incidence of neonatal respiratory distress | 1 day
  Number of neonates needing at least 4 hours of respiratory support with supplemental oxygen, continuous positive airway pressure, or intermittent positive-pressure ventilation during the first 24 hours after delivery.
Incidence of macrosomia | 1 hour
  Number of neonates with birth weight greater than 4000 g or greater than 90% for gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Sinaa Hamdy, MBBCh, Principal Investigator — S Hamdy
Locations (1):
- Ain SHams Maternity Hospital, Cairo, Abbaseya, Egypt